CLINICAL TRIAL: NCT02039986
Title: Effects of Ivacaftor (Kalydeco) Treatment Upon Insulin and Incretin Secretion in Patients With Cystic Fibrosis
Brief Title: Ivacaftor (Kalydeco) and Insulin in Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 13-010465; KELLY13A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation Therapeutics, Inc.)
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Cystic Fibrosis Related Diabetes; Cystic Fibrosis
Keywords: cystic fibrosis; CF; cystic fibrosis related diabetes; CFRD; kalydeco; ivacaftor
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all subjects: all subjects enrolled in same cohort

SUMMARY:
This study is aimed at better understanding the impact of ivacaftor upon insulin and incretin secretion and glucose tolerance in patients with Cystic Fibrosis with a glycine (G551D) mutation. Investigators hypothesize that treatment with ivacaftor improves insulin secretion in individuals with CF.

DETAILED DESCRIPTION:
Cystic Fibrosis Related Diabetes (CFRD) is associated with worse nutritional status, greater pulmonary function decline, and increased mortality, highlighting its relevance in Cystic Fibrosis (CF). CFRD arises primarily from compromised insulin secretion - traditionally considered a by-product of pancreatic exocrine tissue damage and fibrosis. Recent developments in the field of diabetes are propelling a re-examination of this basic explanation. The impact of the cystic fibrosis transmembrane conductance regulator (CFTR) potentiator, ivacaftor, upon insulin secretion and glucose regulation has not been examined, but improved glucose tolerance has been appreciated anecdotally. This study aims to understand the impact of ivacaftor therapy upon blood glucose and insulin and incretin secretion.

ELIGIBILITY:
Inclusion Criteria:

* 6 yrs or older with cystic fibrosis
* at least one G551D CFTR mutation or other non-G551D gating mutation, or residual function CFTR mutation such as, but not limited to, R117H mutation, for which ivacaftor is to be initiated.
* Plan to initiate ivacaftor treatment for FDA approved indications by clinical care team or as part of an ongoing study of ivacaftor for other CFTR mutations, including gating mutations, or residual function mutations.
* not pregnant

Exclusion Criteria:

* established diagnosis of non-CF related diabetes (ie., Type I diabetes)
* history of clinically symptomatic pancreatitis in past year
* prior lung or liver transplant
* severe CF liver disease
* fundoplication-related dumping syndrome
* medical co-morbidities that are not CF-related or are unstable per the Investigator opinion
* acute CF pulmonary exacerbation within 4 weeks prior to study procedures
* treatment with oral or intravenous corticosteroids within 4 weeks of study
* hemoglobin <10g/dL within 90 days of GPA test or at Screening
* abnormal renal function within 90 days of GPA test or at Screening
* long-standing CFRD with fasting hyperglycemia, elevated HbA1C (>8) beyond time surrounding diagnosis of CFRD, significant basal insulin requirement
* inability to perform study specific procedures (MMTT, GPA).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin secretion capacity at 16 weeks | baseline and 16 weeks
  To compare insulin secretion and maximal insulin secretory capacity prior to initiation of ivacaftor and after 16 weeks of ivacaftor treatment in subjects with CF and at least one G551D CFTR mutation, or other CFTR gating mutation, and to explore the impact of ivacaftor upon incretin secretion, incretin regulation of insulin secretion, and glucose excursion during a mixed meal tolerance test in CF.

SECONDARY OUTCOMES:
Composite change from baseline in relationships of insulin secretion and protein and interleukin levels at 16 weeks | baseline and 16 weeks
  To explore the composite relationships of insulin secretion, maximal insulin secretory capacity, and incretin secretion with secreted frizzled protein-4 levels and interleukin 1β levels.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kelly, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States